CLINICAL TRIAL: NCT01292811
Title: Restoration of Upper Limb Function in Individuals With Sub-Acute Spinal Cord Injury
Acronym: MCRCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Financial assistance from agency withdrawn due to financial issues at their end.
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: Rick Hansen Foundation (Other); Ontario Neurotrauma Foundation (Other)
Responsible Party: Principal Investigator, Milos Popovic, Toronto Rehab Chair in Spinal Cord Injury Research, Toronto Rehabilitation Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-048
Record Dates: First submitted 2011-02-07; First posted 2011-02-10 (Estimated); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury; Functional Electrical Stimulation; Hand function; Tetraplegia
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Functional electrical Stimulation (Experimental): The functional electrical stimulation for the treatment group will begin by designing a stimulation protocol that can generate the palmar and/or the lateral grasp on demand. In other words, the stimulation sequence (protocol) will be developed for each patient individually using either Compex Motion or HEWHS stimulator; this will allow the patient, who otherwise cannot grasp, to do so with the system. Both stimulators will be used to deliver the same FES therapy. Stimulation parameters are: 1) balanced, biphasic, current regulated electrical pulses; 2) pulse amplitude from 8 to 50 mA (typical values 17-26 mA); 3) pulse width from 250 to 300 μs; and 4) pulse frequency from 20 to 70 Hz (typical value 25 to 40 Hz).
  Interventions: Device: Functional Electrical Stimulation (Compex Motion Stimulator)
- Control Group (Other): The Control group will receive conventional occupational therapy pertaining to hand function [15].
  The conventional therapy represents control activities against which the FES therapy will be assessed. The conventional occupational therapy includes: a) muscle facilitation exercises emphasizing the neurodevelopmental treatment approach; b) task-specific, repetitive functional training; c) strengthening and motor control training using resistance to available arm motion to increase strength; d) stretching exercises; e) electrical stimulation applied primarily for muscle strengthening (this is not FES but TENS application); f) activities of daily living including self-care where the upper limb was used as an assist if appropriate; and g) caregiver training.
  Interventions: Other: Conventional Occupational therapy

INTERVENTIONS:
Device: Functional Electrical Stimulation (Compex Motion Stimulator) — Functional electrical Stimulation:Parameters of stimulation: 1) balanced, biphasic, current regulated electrical pulses; 2) pulse amplitude from 8 to 50 mA (typical values 17-26 mA); 3) pulse width from250 to 300 μs; and 4) pulse frequency from 20 to 70 Hz (typical value 25 to 40 Hz).
  Other Names: Functional Electrical Stimulation
  Arms: Functional electrical Stimulation
Other: Conventional Occupational therapy — The Control group will receive conventional occupational therapy pertaining to hand function [15].
  The conventional therapy represents control activities against which the FES therapy will be assessed. The conventional occupational therapy includes: a) muscle facilitation exercises emphasizing the neurodevelopmental treatment approach; b) task-specific, repetitive functional training; c) strengthening and motor control training using resistance to available arm motion to increase strength; d) stretching exercises; e) electrical stimulation applied primarily for muscle strengthening (this is not FES but TENS application); f) activities of daily living including self-care where the upper limb was used as an assist if appropriate; and g) caregiver training.
  Arms: Control Group

SUMMARY:
The objective of this research program is to conduct a multi-site clinical randomized control trial that will evaluate the efficacy of functional electrical stimulation based upper limb intervention for people with tetraplegia. This will involve recruiting 84 persons with sub-acute tetraplegia across four sites (Montreal,Toronto, Fredericton and Edmonton) and will serve to evaluate three new Canadian hand function assessments that have been specifically developed for persons with tetraplegia. Although these assessments have been recently tested and have shown considerable promise, further evaluation on their clinical utility (in particular their responsiveness and validity) is required. As well, they need to be compared with one another to determine whether any of these tests is more appropriate for clinical applications or whether further test reduction or augmentation may be required. Having measures that are sensitive and accurate in assessing hand function is key for systematically evaluating emerging therapeutic interventions.

DETAILED DESCRIPTION:
Sustaining a spinal cord injury can impose significant physical dependency and results in financial and psychological challenges to the individual, family and the community at large. For persons with cervical levels of injury (tetraplegia), there is often the loss of hand and upper limb function, which is one of the most devastating consequences of spinal cord injury. The use of hands and upper limbs is needed for daily activities such as feeding, dressing, bathing and toileting. Good hand function plays an important role in the ability to transfer from a bed to a wheelchair, to sit up or to lie down. Not surprisingly, the majority of people with tetraplegia rate recovery of hand function as their highest priority.

One of the most promising approaches to improving hand function is functional electrical stimulation, which uses bursts of short electrical pulses to generate muscle contractions. Functional electrical stimulation enables a person, who would otherwise have paralyzed hands, to grasp and release objects. Although Canadian researchers are at the forefront of upper limb rehabilitation, and have recently developed state-of-the-art therapeutic treatments that involve functional electrical stimulation, there is a strong need to evaluate the efficacy of this intervention. A similar situation also exists with upper limb function assessments. At least three clinically promising upper limb assessments have been recently developed in Canada for individuals with spinal cord injury, which require further evaluation to determine their effectiveness.

The objective of this research program is to conduct a multi-site clinical randomized control trial that will evaluate the efficacy of functional electrical stimulation based upper limb intervention for people with tetraplegia. This will involve recruiting 84 persons with sub-acute tetraplegia across four sites (Montreal,Toronto, Fredericton and Edmonton) and will serve to evaluate three new Canadian hand function assessments that have been specifically developed for persons with tetraplegia. Although these assessments have been recently tested and have shown considerable promise, further evaluation on their clinical utility (in particular their responsiveness and validity) is required. As well, they need to be compared with one another to determine whether any of these tests is more appropriate for clinical applications or whether further test reduction or augmentation may be required. Having measures that are sensitive and accurate in assessing hand function is key for systematically evaluating emerging therapeutic interventions.

The findings of this multi-site clinical trial have the potential to elevate the current standard of upper limb rehabilitation related to hand function by providing higher levels of evidence on the efficacy of functional electrical stimulation therapy intervention. Also, dissemination of the new knowledge gained will translate into better clinical practice since occupational therapists will be able to select better rehabilitation strategies for improving hand function based on solid evidence. By improving the standards of practice, persons with spinal cord injury will have access to a wider range of treatment interventions to restore and improve function in their hands.

ELIGIBILITY:
Inclusion Criteria:

* Sustained a traumatic incomplete SCI between C4 and C7 levels
* 18 years of age or older
* Less than 6 months post injury
* Unable to grasp objects
* Participants must have functional biceps and deltoid muscle strength which allows them to place their hand in the working space in front of themselves, i.e., at least a grade 3 on manual muscle testing
* Participants should have a clear understanding of the goal of the study, which is to compare the FES technology to conventional occupational therapy (which may or may not enhance recovery)
* Participants should be able to read and understand and provide informed consent, and in a situation where there is a difficulty in understanding ( e.g. language barrier), have a relative or friend willing and able to accompany you to all treatment and assessment sessions, for your own safety

Exclusion Criteria:

•Contraindications for FES:

* cardiac pacemakers
* skin lesions, allergy, wound or rash at potential electrode sites
* denervation of targeted muscles
* pressure ulcers
* patient suffers from the cardiovascular conditions such as hypertension that is uncontrolled or autonomic dysreflexia requiring medication
* Patients on Botox therapy for their upper limb or have received Botox for the upper extremity in the last six months
* Participation in any other interventional study that may affect upper extremity function
* Participants with co existing Traumatic brain injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-01; Primary Completion 2014-12-03 (Actual); Study Completion 2014-12-03 (Actual)

PRIMARY OUTCOMES:
Functional Independence Measure to measure burden of care | Change from baseline at 8 weeks and at 6 month follow up
  The FIM is an 18-item ordinal scale, used with all diagnoses within a rehabilitation population. It is viewed as the most useful tool for the assessment of progress during inpatient rehabilitation, and measures independent performance in self-care, sphincter control, transfers, locomotion, communication, and social cognition. By adding the points for each item, the possible total score ranges from 18 (lowest) to 126 (highest) level of independence

SECONDARY OUTCOMES:
Graded Redefined Assessment of Strength Sensibility and Prehension to assess gross motor function and sensation of the hand | Change from basline upon completion of therapy (8 weeks)and at 6 month follow
  This test combines the features of several other tests that have been used to assess hand and upper limb function in the peripheral hand population. The key features of the GRASSP are: 1) measures each of the sensory, motor and grasping capabilities
Jamar® Hydraulic Hand Dynamometer to measure grip and pinch force | Change from Baseline at 8 weeks and 6 months
  Jamar® Hydraulic Hand Dynamometer will be used to measure isometric grip force. The range of the sensor is from 0 to 90 kg.
Action Research Arm Test to measure upper extremity function | Change from Baseline at 8 weeks and 6 months
  measure upper extremity function
Toronto Rehab Hand Function Test (TR-HFT)to measure gross motor hand function | Change from Baseline at 8 weeks and 6 months
  measure gross motor hand function
REJOYCE | Change from Baseline at 8 weeks and 6 months
  to measure change in upper extremity range of motion and various grip strengths
Spinal Cord Independence Measure | Change from Baseline at 8 weeks and 6 months
  to measure impairment

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Milos R Popovic, PhD, Principal Investigator — Toronto Rehabilitation Institute
Locations (1):
- Toronto Rehabilitation Institute, Toronto, Ontario, Canada